CLINICAL TRIAL: NCT05292118
Title: Navitian Post-Market Clinical Follow-up Study
Brief Title: Navitian PMCF Study ( rEPIC04C )
Acronym: rEPIC04C
Status: Completed | Type: Observational
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Other Study IDs: Navitian PMCF Study
Record Dates: First submitted 2022-03-14; First posted 2022-03-23 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2024-08

CONDITIONS: Coronary Artery Disease (CAD); Ischemic Heart Disease
Keywords: MDR (Medical Device Regulations); PMCF (Post-Market Clinical Follow-up); Coronary microcatheter
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Coronary Artery Disease (CAD)
  Interventions: Device: Navitian

INTERVENTIONS:
Device: Navitian — Patients in whom treatment with (Navitian) has been attempted

SUMMARY:
Multicenter, prospective, non-randomized, post-market clinical follow-up (PMCF) study to confirm and support the clinical safety and performance of Navitian to meet EU Medical Device regulation (MDR) requirements in all the CONSECUTIVE patients treated with Navitian.

DETAILED DESCRIPTION:
The objective of this multicenter, prospective, non-randomized, post-market clinical follow-up (PMCF) study is to confirm and support the clinical safety and performance of the Navitian in a NON-SELECTED, Real World population under daily clinical practice when used as intended by the manufacturer to meet EU Medical Device regulation requirements for post-market clinical follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient treated with Navitian according to routine hospital practice and following instructions for use
* Informed consent signed

Exclusion Criteria:

* Not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with Navitian according to routine hospital practice and following instructions for use
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2024-07-11 (Actual); Study Completion 2024-07-11 (Actual)

PRIMARY OUTCOMES:
Safety Endpoint. Freedom fromTarget Lesion Failure | 7 days
  Freedom from TARGET LESION FAILURE (TLF), composite endpoint of Cardiac death, Myocardial infarction, and new Target Lesion Revascularization (TLR).

SECONDARY OUTCOMES:
Efficacy Endpoint. Freedom from Target Lesion Failure | 7 days
  Freedom from TARGET LESION FAILURE (TLF), composite endpoint of Cardiac death, Myocardial infarction, and new Target Lesion Revascularization (TLR).
Freedom from Device rupture | During percutaneous coronary intervention (PCI)
  Freedom from Device rupture
Freedom from Kinking | During PCI
  Freedom from Kinking
Freedom from Complicated withdrawal | During PCI
  Freedom from Complicated withdrawal
Freedom from Coronary perforation | During PCI
  Freedom from Coronary perforation
Freedom from Coronary dissection >C | During PCI
  Freedom from Coronary dissection >C
Freedom from No reflow | During PCI
  Freedom from No reflow
Freedom from Coronary thrombosis | During PCI
  Freedom from Coronary thrombosis

CONTACTS AND LOCATIONS:
Locations (8):
- Centro Hospitalar Vila Nova de Gaia, Vila Nova de Gaia, Portugal
- Spain (7):
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Juan Ramon Jimenez, Huelva
  - Hospital Universitario de Leon, León
  - Hospital Universitario Lucus Agusti, Lugo
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Clinico Universitario de Valladolid, Valladolid

REFERENCES:
- [Background] Gruntzig A. Transluminal dilatation of coronary-artery stenosis. Lancet. 1978 Feb 4;1(8058):263. doi: 10.1016/s0140-6736(78)90500-7. No abstract available. PMID 74678
- [Background] Obata JE, Nakamura T, Kitta Y, Saito Y, Sano K, Fujioka D, Kawabata K, Kugiyama K. Usefulness of a collateral channel dilator for antegrade treatment of chronic total occlusion of a coronary artery. J Interv Cardiol. 2012 Dec;25(6):533-9. doi: 10.1111/j.1540-8183.2012.00758.x. Epub 2012 Jul 23. PMID 22823494